CLINICAL TRIAL: NCT05450692
Title: A Phase III, Open-label, Randomised, Multicentre Study of Ceralasertib Plus Durvalumab Versus Docetaxel in Patients With Advanced or Metastatic Non-Small Cell Lung Cancer Without Actionable Genomic Alterations, and Whose Disease Has Progressed On or After Prior Anti-PD-(L)1 Therapy and Platinum-based Chemotherapy: LATIFY
Brief Title: A Phase III Study of Ceralasertib Plus Durvalumab Versus Docetaxel in Patients With Non Small Cell Lung Cancer (NSCLC) Whose Disease Progressed On or After Prior Anti PD (L)1 Therapy And Platinum Based Chemotherapy
Acronym: LATIFY
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Parexel (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D533BC00001; 2022-000493-26 (EudraCT Number)
Record Dates: First submitted 2022-07-06; First posted 2022-07-11 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Advanced or Metastatic Non-Small Cell Lung Cancer
Keywords: Durvalumab; Ceralasertib; Docetaxel; Lung cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms | interventions — ceralasertib; durvalumab; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Group A: Ceralasertib plus durvalumab combination therapy (Experimental): Participants will be administered ceralasertib orally followed by durvalumab administered intravenously.
  Interventions: Drug: Ceralasertib; Drug: Durvalumab
- Group B: Docetaxel monotherapy (Active Comparator): Participants will be administered docetaxel (standard of care) administered intravenously.
  Interventions: Drug: Docetaxel

INTERVENTIONS:
Drug: Ceralasertib — Participants will receive ceralasertib oral tablets.
  Arms: Group A: Ceralasertib plus durvalumab combination therapy
Drug: Durvalumab — Participants will receive durvalumab as an intravenous infusion.
  Arms: Group A: Ceralasertib plus durvalumab combination therapy
Drug: Docetaxel — Participants will received docetaxel as an intravenous infusion.
  Arms: Group B: Docetaxel monotherapy

SUMMARY:
This study will assess the efficacy and safety of the combination of ceralasertib and durvalumab versus standard of care docetaxel in patients with locally advanced and metastatic NSCLC after progression on prior anti-PD-(L)1 therapy and platinum-based chemotherapy.

DETAILED DESCRIPTION:
This study will consist of two treatment arms (Groups A and B).

Participants will be randomised in a 1:1 ratio to one of the two treatment groups:

* Group A: Ceralasertib plus durvalumab combination therapy Each 28-day cycle will begin with ceralasertib administered orally followed by durvalumab administered intravenously.
* Group B: Docetaxel monotherapy Each 21-day cycle will begin with the administration of docetaxel.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically documented NSCLC that is locally advanced or metastatic according to Version 8 of the IASLC Staging Manual in Thoracic Oncology.
* Documented epidermal growth receptor factor (EGFR) and anaplastic lymphoma kinase (ALK) wild-type status as determined at a local laboratory.
* Documented radiological PD whilst on or after receiving the most recent treatment regimen.
* Eligible for second- or third-line therapy and must have received an anti-PD-(L)1 therapy and a platinum doublet containing therapy for locally advanced or metastatic NSCLC either separately or in combination.
* Eastern Cooperative Oncology Group (ECOG)/World Health Organization (WHO) performance status of 0 or 1.
* Adequate organ function and marrow reserve
* Minimum life expectancy of 12 weeks.
* Body weight > 30 kg and no cancer-associated cachexia.
* Negative pregnancy test (serum test) for women of childbearing potential (WOCBP).

Exclusion Criteria:

* Participant with mixed SCLC and NSCLC histology.
* History of another primary malignancy except for malignancy treated with curative intent with no known active disease ≥ 5 years before the first dose of study intervention.
* Persistent toxicities (CTCAE Grade > 2) caused by previous anticancer therapy.
* Active or prior documented autoimmune or inflammatory disorders.
* Participants who have received more than one line of prior anti-PD-(L)1, either alone or in any combination.
* Participants:

  1. Must not have experienced a toxicity that led to permanent discontinuation of the prior anti-PD(L)1 therapy.
  2. All AEs while receiving prior anti-PD(L)1 therapy must have completely resolved.
  3. Must not have experienced a Grade ≥ 3 immune-mediated adverse event (imAE) or an immune-related neurologic or ocular AE of any grade while receiving prior anti-PD(L)1 therapy.
  4. Must not have required the use of additional immunosuppression other than corticosteroids for the management of an AE, not have experienced recurrence of an AE if re-challenged, and not currently require maintenance doses of > 10 mg prednisone or equivalent per day.
* Participants who have received more than one prior line of platinum-based chemotherapy in metastatic setting.
* Participants who have received a prior ataxia telangiectasia and Rad3-related protein (ATR) inhibitor.

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 594 (Actual)
Dates: Start 2022-09-15 (Actual); Primary Completion 2025-10-06 (Actual); Study Completion 2026-10-30 (Estimated)

PRIMARY OUTCOMES:
Overall Survival (OS) | Every 3 months (± 1 week) following objective progression of disease (PD) or treatment discontinuation (up to three years)
  The superiority of ceralasertib plus durvalumab combination therapy relative to docetaxel will be demonstrated by assessment of OS (HR with 95% CI and p-value) in participants with advanced NSCLC after second- or third-line therapy and without actionable genomic alterations. OS is defined as time from randomisation until the date of death due to any cause.

SECONDARY OUTCOMES:
Progression-Free Survival (PFS) | Up to 3 years
  PFS will be defined as the time from the date of randomisation until the date of objective PD.
Objective Response Rate (ORR) | Up to 3 years
  ORR is defined as the proportion of participant who have a Complete Response (CR) or Partial Response (PR) per RECIST 1.1.
Duration of Response (DoR) | Up to 3 years
  DoR is defined as the time from the date of first documented response until date of documented progression per RECIST 1.1.
Time To Response (TTR) | Up to 3 years
  TTR is defined as the time from randomisation until the date of first documented objective response.
Disease Control Rate (DCR) | At Week 18
  DCR at 18 weeks is defined as the percentage of participants who have a CR or PR or who have stable disease (SD) for at least 17 weeks.
Time to second progression or death (PFS2) | Up to 3 years
  Time from randomisation to PFS2 will be defined as the time from the randomisation to the earliest of the progression event (following the initial progression), subsequent to first subsequent therapy or death.
Overall Survival (OS) at 12 months | At 12 months
  OS is defined as time from randomisation until the data of death due to any cause.
Time To Deterioration (TTD) of health-related quality of life (QoL) | Up to 3 years
  TTD is defined as the time from randomisation until the date of first confirmed deterioration.
TTD of physical function | Up to 3 years
  TTD in physical functioning is measured by the EORTC QLQ-C30 Physical Function subscale of the EORTC QLQ-C30.
Plasma concentrations for ceralasertib plus durvalumab combination therapy | Up to 3 years
  The PK plasma concentration of ceralasertib when administered in combination with durvalumab will be assessed.
Number of participants with Adverse Evens (AEs) | Up to 3 years
  The safety and tolerability of ceralasertib plus durvalumab combination therapy as compared with docetaxel will be assessed.

CONTACTS AND LOCATIONS:
Locations (169):
- United States (28):
  - Research Site, Mobile, Alabama
  - Research Site, Chandler, Arizona
  - Research Site, Los Alamitos, California
  - Research Site, Los Angeles, California
  - Research Site, Whittier, California
  - Research Site, Jacksonville, Florida
  - Research Site, Orlando, Florida
  - Research Site, Tampa, Florida
  - Research Site, Athens, Georgia
  - Research Site, Atlanta, Georgia
  - Research Site, Fort Wayne, Indiana
  - Research Site, Baltimore, Maryland
  - Research Site, Bethesda, Maryland
  - Research Site, Rockville, Maryland
  - Research Site, Hattiesburg, Mississippi
  - Research Site, St Louis, Missouri
  - Research Site, Omaha, Nebraska
  - Research Site, Reno, Nevada
  - Research Site, Charlotte, North Carolina
  - Research Site, Winston-Salem, North Carolina
  - Research Site, Canton, Ohio
  - Research Site, Cleveland, Ohio
  - Research Site, Allentown, Pennsylvania
  - Research Site, York, Pennsylvania
  - Research Site, Houston, Texas
  - Research Site, Huntsville, Texas
  - Research Site, Kingwood, Texas
  - Research Site, Appleton, Wisconsin
- Argentina (4):
  - Research Site, Buenos Aires
  - Research Site, Pergamino
  - Research Site, Rosario
  - Research Site, San Juan
- Australia (5):
  - Research Site, Elizabeth Vale
  - Research Site, Lismore
  - Research Site, Murdoch
  - Research Site, South Brisbane
  - Research Site, Wollongong
- Belgium (4):
  - Research Site, Charleroi
  - Research Site, Ghent
  - Research Site, Libramont-Chevigny
  - Research Site, Roeselare
- Brazil (4):
  - Research Site, Fortaleza
  - Research Site, Porto Alegre
  - Research Site, Salvador
  - Research Site, São Paulo
- Canada (6):
  - Research Site, Vancouver, British Columbia
  - Research Site, Newmarket, Ontario
  - Research Site, Chicoutimi, Quebec
  - Research Site, Montreal, Quebec
  - Research Site, Québec, Quebec
  - Research Site, Rimouski, Quebec
- China (20):
  - Research Site, Baoding
  - Research Site, Beijing
  - Research Site, Changsha
  - Research Site, Chengdu
  - Research Site, Deyang
  - Research Site, Guangzhou
  - Research Site, Hangzhou
  - Research Site, Hefei
  - Research Site, Jinan
  - Research Site, Linyi
  - Research Site, Nanchang
  - Research Site, Nanjing
  - Research Site, Nanning
  - Research Site, Nashik
  - Research Site, Qingdao
  - Research Site, Taiyuan
  - Research Site, Tianjin
  - Research Site, Wuhan
  - Research Site, Zhanjiang
  - Research Site, Zhengzhou
- France (14):
  - Research Site, Angers
  - Research Site, Clamart
  - Research Site, Clermont-Ferrand
  - Research Site, Créteil
  - Research Site, Lyon
  - Research Site, Montpellier
  - Research Site, Nantes
  - Research Site, Paris
  - Research Site, Pessac
  - Research Site, Saint-Herblain
  - Research Site, Saint-Quentin
  - Research Site, Vantoux
  - Research Site, Villefranche-sur-Saône
  - Research Site, Villejuif
- Germany (7):
  - Research Site, Berlin
  - Research Site, Freiburg im Breisgau
  - Research Site, Gauting
  - Research Site, Karlsruhe
  - Research Site, Kempten
  - Research Site, Löwenstein
  - Research Site, Moers
- Hong Kong (3):
  - Research Site, Hong Kong
  - Research Site, King's Park
  - Research Site, Tun Mun
- Hungary (2):
  - Research Site, Budapest
  - Research Site, Székesfehérvár
- India (3):
  - Research Site, Jaipur
  - Research Site, Pune
  - Research Site, Surat
- Ireland (3):
  - Research Site, Cork
  - Research Site, Dublin
  - Research Site, Limerick
- Italy (12):
  - Research Site, Aviano
  - Research Site, Livorno
  - Research Site, Meldola
  - Research Site, Milan
  - Research Site, Monza
  - Research Site, Napoli
  - Research Site, Padua
  - Research Site, Parma
  - Research Site, Perugia
  - Research Site, Roma
  - Research Site, Rozzano
  - Research Site, Verona
- Japan (15):
  - Research Site, Bunkyō City
  - Research Site, Chūōku
  - Research Site, Kōtoku
  - Research Site, Kurashiki-shi
  - Research Site, Kurume-shi
  - Research Site, Matsuyama
  - Research Site, Nagoya
  - Research Site, Niigata
  - Research Site, Osaka
  - Research Site, Sakaishi
  - Research Site, Sapporo
  - Research Site, Sendai
  - Research Site, Sunto-gun
  - Research Site, Toyoake-shi
  - Research Site, Yokohama
- Netherlands (2):
  - Research Site, Heerlen
  - Research Site, Tilburg
- Poland (4):
  - Research Site, Gdansk
  - Research Site, Krakow
  - Research Site, Poznan
  - Research Site, Skórzewo
- Romania (6):
  - Research Site, Bucharest
  - Research Site, Cluj-Napoca
  - Research Site, Craiova
  - Research Site, Floreşti
  - Research Site, Oradea
  - Research Site, Timișoara
- Research Site, Belgrade, Serbia
- South Korea (3):
  - Research Site, Cheongju-si
  - Research Site, Seoul
  - Research Site, Suwon
- Spain (14):
  - Research Site, A Coruña
  - Research Site, Barcelona
  - Research Site, Castellon
  - Research Site, Córdoba
  - Research Site, Hospitalet deLlobregat
  - Research Site, Madrid
  - Research Site, Málaga
  - Research Site, Ourense
  - Research Site, Palma de Mallorca
  - Research Site, Pamplona
  - Research Site, Pozuelo de Alarcón
  - Research Site, Sabadell
  - Research Site, Servilla
  - Research Site, Zaragoza
- Taiwan (5):
  - Research Site, Taichung
  - Research Site, Tainan
  - Research Site, Taipei
  - Research Site, Taoyuan District
  - Research Site, Yunlin
- United Kingdom (4):
  - Research Site, Guildford
  - Research Site, Metropolitan Borough of Wirral
  - Research Site, Stevenage
  - Research Site, Sutton

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the deidentified individual patient-level data in an approved sponsored tool. Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- See also: Lung Cancer Study Locator details (for US) — https://www.lungcancerstudylocator.com/trial/listing/350218